CLINICAL TRIAL: NCT00953472
Title: Clinical Proteomics and Protein Therapeutics in Human Hypertension (BNP in Human Hypertension - Phase 1)
Brief Title: B-type Natriuretic Peptide (BNP) in Human Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-003032; MC cardiorenal lab funds
Record Dates: First submitted 2009-04-02; First posted 2009-08-06 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension Stage 1
Keywords: hypertension treatment
MeSH Terms: conditions — Hypertension | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: brain natriuretic peptide — start 10 mcg/kg (2 participants), 7 mcg/kg (2 participants), 5 mcg/kg (2 participants) and 2 mcg/kg (2 participants)
Other: no-added salt diet — instruction to reduce salt for one week prior to study

SUMMARY:
The investigators working hypothesis is that human hypertension is in part due to a derangement in the endocrine function of the heart - a primary or secondary mechanism - resulting in a relative deficiency of the natriuretic peptides (NP). The remodeled hypertensive heart could result in altered processing and degradation of B-type NP resulting in altered molecular forms with decreased biological activity. The investigators further hypothesized the chronic administration of BNP in subjects with hypertension, is feasible, safe and will induce a sustained reduction in blood pressure.

DETAILED DESCRIPTION:
Ongoing investigations by our laboratory group and others have established that the heart is an endocrine organ as well as a pump. The heart synthesizes and secretes two peptide hormones - atrial natriuretic peptide (ANP) and B-type natriuretic peptide (BNP) - that are endogenous ligands for a particulate guanylyl cyclase receptor (NPR-A). Following receptor binding and generation of its second messenger cGMP, the natriuretic peptides (NPs) mediate biological actions which include natriuresis, inhibition of the renin-angiotensin system and vasodilatation with local autocrine and paracrine actions in the heart to include inhibition of fibrosis and enhancement of diastolic function.

Hypertension remains a global burden in cardiovascular disease leading to stroke, myocardial infarction and heart failure. Its myocardial complications result from increased mechanical load on the heart. Under physiological conditions of increased myocardial load and resulting myocardial stretch, ANP and BNP synthesis and secretion occur contributing to maintenance of optimal cardiorenal and blood pressure homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Subjects with stage 1 hypertension (SBP: 140-159 mm Hg or DBP 90-99 mm Hg) If on therapy, it must be stable for at least 1 month.

Exclusion Criteria:

* Congestive Heart Failure (any NYHA class).
* EF < 50%.
* Myocardial infarction within 3 months of screening.
* Unstable angina within 14 days of screening, or any evidence of myocardial ischemia.
* Moderate to severe pulmonary hypertension.
* Valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis.
* Sustained VT or V-fib within 14 days of screening.
* Sustained Atrial Fibrillation.
* Second or third degree AV block without a permanent cardiac pacemaker.
* CVA within 3 months of screening, or other evidence of significantly compromised CNS perfusion.
* Total bilirubin of >1.5 mg/dL or AST and ALT 1.5 times the upper limit of normal range.
* Renal insufficiency assessed by calculated GFR < 60 ml/min (Cockroft-Gault equation).
* Serum sodium of < 125 mEq/dL or > 160 mEq/dL.
* Serum potassium of < 3.5 mEq/dL or > 5.0 mEq/dL.
* Women taking hormonal contraceptives.
* Body Mass Index (BMI) > 35.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The blood pressure will decrease with BNP injections | during study intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States